CLINICAL TRIAL: NCT04718012
Title: Retrospective, Observational, Multi-center Study Evaluating the Efficacy and Tolerance of Brigatinib in the Management of Rearranged CBNPC ROS1
Acronym: BRIGAROS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: BRIGAROS
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Lung Cancer ROS Translocated
Keywords: Brigatinib, lung cancer, ROS1
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ROS1 translocated Non small cell lung cancer (NSCLC) is a rare type of lung cancer with few datas. We collected datas concerning patients with ROS1 translocated NSCLC who received Brigatinib in the Compassionate Access after two others Tyrosine kinase Inhibitors

DETAILED DESCRIPTION:
Lung cancer is the most common cancer worldwide and the leading cause of cancer death in Western countries. Non-small cell lung cancer (NSCLC) is the most usual form (80-85%) of lung cancers. Unfortunately, at the time of diagnosis, most patients present with metastatic or advanced disease. Significant advances have been made in recent years on knowledge of oncogenesis of NSCLC in particularly the discovery of specific oncogenic drivers playing key role in oncogenic addiction responsible for the occurrence of NSCLC.

ROS1 translocation is found in1 to 2 % of non small cell lung cancer. Due to this rare subtype of cancer, we have few datas. ROS1 translocation is found in a rather younger population, with a predominance of woman and non smoker. ROS1 translocation can be detected by immunohistochemistry and confirmed by FISH or RNA fusion technics.

Crizotinib demonstrated his interest in the phase 1 trial PROFILE 1001 with an objective response rate of 72% tested on 52 patients, the median progression free survival was 19,3 months, overall survival of 51% at 48 months.

Similar datas were found in different cohortes. A chinese study of 23 patients receiving crizotinib, the objective response rate was 56,5%, a median progression free survival of 14,5 months. A european retrospective cohorte EUROS1 of 30 patients receiving crizotinib found a progression free survival of 9,1 months, an objective response rate of 80% . A prospective european study EUCROSS included 34 patients with an objective response rate of 70% and a progression free survival of 20 months. The Acsé crizotinib cohorte included 37 patients ROS1 translocated, the objective response rate was lower at 47,2% in this study with heavily pretreated population.

Ceritinib has been studied in a phase 2 study of 32 patients in whom 30 patients where treatment naifs of crizotinib, the objective response rate was 62%.

Lorlatinib was studied in a phase1-2 trial, including 69 ROS1 patients, 21 were TKI naifs, 40 pretreated with crizotinib and 8 treated with one or two others TKI, with objective response rate of 62% in the naive population, and 41% on the entire cohorte.

More recently, Entrectinib demonstrated his interest in a pooled study of 3 trial, 53 patients were ROS1 translocated and had an objective response rate of 77% with this new molecule.

Few datas are available about brigatinib in ROS1 translocated patients, only three patients ROS1 were included in the brigatinib phase 1 trial. The aim of this study is to obtain more datas of efficacy, safety, among patients receiving Brigatinib with the compationnate access in France

ELIGIBILITY:
Inclusion Criteria:

* patient with CBNPC transloated ROS1
* Treatment by Brigatinib as part of compassionate access in France
* Patient > 18 years old

Exclusion Criteria:

* Refusal of the patient to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CBNPC when they visit the respiratory ward
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2021-10-17 (Actual); Study Completion 2021-10-17 (Actual)

PRIMARY OUTCOMES:
progression-free survival on Brigatinib in patients with ROS1 translocated CBNPCtransloated CBNPC | 27 months

SECONDARY OUTCOMES:
overall survival | 27 months
Number of side effects associated with brigatinib | 27 months
Types of side efects associated with brigatinib | 27 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHI Créteil, Créteil, France